CLINICAL TRIAL: NCT03377049
Title: C-arm Cone Beam CTA and CTP With Acetazolamide Challenge in Aneurysmal Subarachnoid Hemorrhage: Evaluating Predictability for Early Ischemia in Cerebral Vasospasm
Brief Title: Acetazolamide Challenge With Perfusion in the Prediction of Cerebral Vasospasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-1510; SMPH/NEURO SURG/NEURO SURG (Other: UW Madison); A535700 (Other: UW Madison); Protocol Version 4/28/2020 (Other: UW Madison)
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Vasospasm, Cerebral
Keywords: acetazolamide challenge; cerebral vasospasm; aneurysmal subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Acetazolamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acetazolamide Challenge (Experimental): Participants entered into the study as a cohort, will because of their participation, undergo only two additional digital subtraction angiogram (DSA) imaging acquisitions. These will be done in conjunction with their standard diagnostic DSA evaluation and consist of two CBCTPs, one before and one after administration of 1 g acetazolamide through a peripheral IV line. Each CBCTP will require administration of 75-100 mL iodinated contrast medium also through an intravenous line. Neither of these imaging studies will be used for clinical decision making, but would be processed and evaluated at later date for a formal analysis of the results. Following completion of diagnostic imaging subjects will receive the usual standard of care for treatment of their ruptured aneurysm i.e. endovascular embolization or open surgical clipping.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — 1 g acetazolamide through a peripheral IV line
  Other Names: Diamox

SUMMARY:
The investigators propose a technique using cone beam CT perfusion (CBCTP) imaging with an acetazolamide challenge as a potential diagnostic tool to detect a defect in cerebral autoregulation at a time when it has not yet caused clinically apparent signs or symptoms. 30 participants will be enrolled at the University of Wisconsin - Madison and can expect to be on study for about 2 weeks.

DETAILED DESCRIPTION:
Acetazolamide or vasodilatory challenge should identify subjects having a abnormal cerebrovascular reactivity capacity. More specifically, after receiving the drug there will not be the expected increase in cerebral blood flow (CBF) in some of the subjects because they are already suffering from a disturbance in the vasculature's ability to respond to the signal for vasodilation. The investigators believe the presence of this deficit will be helpful in identifying patients who are at risk for potential brain ischemia due to this decreased capacity to autoregulate if/when clinically significant vasospasm occurs. The investigators predict that acetazolamide-activated regional cerebral blood flow studies will be more sensitive in the detection of mild cerebral vasospasm and will not just detect changes in cerebral blood flow as does standard perfusion imaging, but will provide information regarding changes in cerebrovascular reactivity. Under these circumstances, a better predictor of those patients at risk of cerebral infarction due to delayed vasospasm would be delineated. Identifying this "high-risk cohort" prior to the onset of clinically apparent symptoms would result in the institution of preventative measures such as triple H therapy.

The objective of this proposal is to conduct a feasibility study of acetazolamide activated C-arm cone beam CT perfusion (CBCTP) to determine its application in the prediction of symptomatic cerebral vasospasm (i.e. ischemia or stroke) in patients with aneurysmal subarachnoid hemorrhage. The initial plan is to obtain C-arm CBCTP pre- and post-intravenous infusion of 1g acetazolamide within 24 hours of symptom onset in aneurysmal subarachnoid hemorrhage patients. The hypothesis is that some of these patients that will later develop clinical vasospasm of a degree sufficient to cause cerebral ischemia. The investigators believe this cohort of patients will demonstrate altered cerebrovascular reactivity during the acetazolamide challenge at a time before there is either angiographic evidence of vasospasm or clinical evidence of abnormal perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aneurysmal subarachnoid hemorrhage presenting to our institution within 24 hours of symptom onset
* Adults, 18 years of age or older
* Women of childbearing potential must not be pregnant (negative urine pregnancy test)

Exclusion Criteria:

* Contraindication to acetazolamide (i.e. sulfonamide allergy, renal or liver failure)
* Contraindication to contrast media (Allergy or abnormal serum Cr and/or GFR based on current UW guidelines for IV contrast)
* Renal insufficiency, history of renal failure or renal transplant
* Hunt and Hess grade 1 and 5 (Attached protocol provides details on the grading scale. Grade 1 have lowest yield for vasospasm and Grade 5 are by definition critically ill and unstable patients)
* Critically ill patients who are unstable and who cannot undergo scans within the proposed timeline i.e. within 24 hours of the onset of their symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azam Ahmed, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shinoda J, Kimura T, Funakoshi T, Araki Y, Imao Y. Acetazolamide reactivity on cerebral blood flow in patients with subarachnoid haemorrhage. Acta Neurochir (Wien). 1991;109(3-4):102-8. doi: 10.1007/BF01403003. PMID 1858527
- [Background] Tanaka A, Yoshinaga S, Nakayama Y, Tomonaga M. Cerebral blood flow and the response to acetazolamide during the acute, subacute, and chronic stages of aneurysmal subarachnoid hemorrhage. Neurol Med Chir (Tokyo). 1998 Oct;38(10):623-30; discussion 630-2. doi: 10.2176/nmc.38.623. PMID 9861845
- [Background] Lee KH, Lukovits T, Friedman JA. "Triple-H" therapy for cerebral vasospasm following subarachnoid hemorrhage. Neurocrit Care. 2006;4(1):68-76. doi: 10.1385/NCC:4:1:068. PMID 16498198
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Sullivan HG, Kingsbury TB 4th, Morgan ME, Jeffcoat RD, Allison JD, Goode JJ, McDonnell DE. The rCBF response to Diamox in normal subjects and cerebrovascular disease patients. J Neurosurg. 1987 Oct;67(4):525-34. doi: 10.3171/jns.1987.67.4.0525. PMID 3655890
- [Background] Hinson JS, Ehmann MR, Fine DM, Fishman EK, Toerper MF, Rothman RE, Klein EY. Risk of Acute Kidney Injury After Intravenous Contrast Media Administration. Ann Emerg Med. 2017 May;69(5):577-586.e4. doi: 10.1016/j.annemergmed.2016.11.021. Epub 2017 Jan 25. PMID 28131489
- [Background] Hauge A, Nicolaysen G, Thoresen M. Acute effects of acetazolamide on cerebral blood flow in man. Acta Physiol Scand. 1983 Feb;117(2):233-9. doi: 10.1111/j.1748-1716.1983.tb07202.x. PMID 6869033
- [Background] Kimura T, Shinoda J, Funakoshi T. Prediction of cerebral infarction due to vasospasm following aneurysmal subarachnoid haemorrhage using acetazolamide-activated 123I-IMP SPECT. Acta Neurochir (Wien). 1993;123(3-4):125-8. doi: 10.1007/BF01401867. PMID 8237489
- [Background] Bruce RJ, Djamali A, Shinki K, Michel SJ, Fine JP, Pozniak MA. Background fluctuation of kidney function versus contrast-induced nephrotoxicity. AJR Am J Roentgenol. 2009 Mar;192(3):711-8. doi: 10.2214/AJR.08.1413. PMID 19234268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 2019 to April 2022.
Period: Overall Study
Arm/Group | Acetazolamide Challenge
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acetazolamide Challenge
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2
  40-49 years | 0
  50-59 years | 3
  60-69 years | 3
  70-79 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Delayed Cerebral Vasospasm
Description: Clinical neurological deterioration not attributable to other causes, mores specifically not due to re-bleeding, hydrocephalus, or metabolic changes.
Time Frame: Day 1-14 during the hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide Challenge
Number analyzed (Participants) | 11
Participants | 2

2. Secondary Outcome: Relative Percent Change in Cerebral Blood Flow
Description: The data that will be statistically compared is the pre-diamox perfusion in comparison to the post-diamox perfusion. A statistically significant change increase in CBF represents an appropriate response to Diamox. Lack of change in CBF or decrease in CBF could be suggestive of potential for developing vasospasm.
Time Frame: pre and post perfusion during imaging procedure, up to an hour
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acetazolamide Challenge
Number analyzed (Participants) | 11
percent change | 20.722 (13.967)

3. Secondary Outcome: Percent Change in Left Hemisphere Brain Imaging Maps
Description: Using perfusion map values, relative percent change will be calculated
Time Frame: pre and post perfusion during imaging procedure, up to an hour
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acetazolamide Challenge
Number analyzed (Participants) | 11
percent change | 19.785 (13.488)

4. Secondary Outcome: Percent Change in Right Hemisphere Brain Imaging Maps
Description: Using perfusion map values, relative percent change will be calculated
Time Frame: pre and post perfusion during imaging procedure, up to an hour
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acetazolamide Challenge
Number analyzed (Participants) | 11
percent change | 21.659 (15.046)

ADVERSE EVENTS:
Time Frame: Days 1-14 during hospitalization
Arm/Group | Acetazolamide Challenge
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide Challenge (N=11)
Cardiomyopathy (Cardiac disorders) | 1 (1)
External Ventricular Drainage infection (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide Challenge (N=11)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT03377049/Prot_SAP_000.pdf